CLINICAL TRIAL: NCT02493400
Title: Physiotherapist Led Group-exercise Compared Physical Activity on Prescription in Older Patients With Atrial Fibrillation, a 3 Months Follow-up
Brief Title: Physiotherapist Led Group-exercise Compared Physical Activity on Prescription, a 3 Months Follow-up
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: Goteborg follow up flimmer
Record Dates: First submitted 2015-07-06; First posted 2015-07-09 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Atrial Fibrillation
Keywords: Follow up; Exercise; Rehabilitation
MeSH Terms: conditions — Atrial Fibrillation; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Exercise group: A follow up from 3 months detraining from the exercise group. Patients follows their earlier randomisation.
  Interventions: Other: No intervention in the follow up study.
- Active Comparator: PAP group: A follow up from 3 months detraining from the active comparator group. Patients follows their earlier randomisation.
  Interventions: Other: No intervention in the follow up study.

INTERVENTIONS:
Other: No intervention in the follow up study.

SUMMARY:
To investigate the effect of exercise or PAP prescription 3 months after completion of the study "Should elderly patients with atrial fibrillation be offered physiotherapist group exercise or can physical activity on prescription (PAP) be used as an alternative?" regarding level of physical fitness, physical activity, heart rate and health related quality of life (HR-QoL). Also if any of the investigated variables can predict the possible change in physical fitness.

DETAILED DESCRIPTION:
Patients who have completed study will be offered a follow-up after 3 months regarding physical fitness, physical activity, heart rate and HR-QoL. Physical fitness will be measured by a symptom limited bicycle test and a muscle endurance test. Physical activity will be measured by accelerometer and the International Physical Activity Questionnaire (IPAQ) and a physical activity diary, HR-QoL will be measured by short form (SF-36).

ELIGIBILITY:
Inclusion Criteria:

* Completed the study "Should elderly patients with atrial fibrillation be offered physiotherapist group exercise or can physical activity on prescription (PAP) be used as an alternative?"

Exclusion Criteria:

* Not completed the above study or denied participation in follow up

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients who have completed the primary study will be offered a follow-up after 3 months
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2014-08; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Physical fitness | 3 months follow up
  Working capacity in watt

SECONDARY OUTCOMES:
Physical activity | 3 months follow up
  accelerometer and questionnaire
Health related quality of life | 3 months follow up
  questionnaire short form (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Asa Cider, Phd RPT, Study Director — Institute of Neuroscience and Physiology/Physiotherapy
Locations (1):
- Sahlgrenska university hospital and Alingsås hospital, Gothenburg, Sweden